CLINICAL TRIAL: NCT02126800
Title: Rapid Medical Donation Programme for Breast Cancer to Examine Tumour Heterogeneity
Brief Title: Rapid Medical Donation Programme for Breast Cancer
Acronym: LEGACY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Breakthrough Breast Cancer (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3995
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metastatic breast cancer
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Treatment of breast cancer has traditionally been based on the primary tumour's features in the breast. Only recently, when cancer returns at other sites, has there been an attempt to biopsy the metastatic disease and change treatments accordingly. A 'repeat biopsy' can be technically difficult, painful and, when possible, only represents a small sample of one of many metastases.

Even when one deposit responds to a new treatment, a neighbouring one may continue to grow. There is an urgent need to characterise all deposits, particularly the lethal ones which progress despite all treatments.

This study will enable the comprehensive analysis of the metastatic process and the evolution of the breast cancer through the course of its treatment. Patients who have consented during life to donate their tissues for molecular analysis will provide the means for such an analysis.

Main aims:

* To comprehensively and systematically examine metastatic breast cancer by its detailed exploratory molecular characterization to elucidate the possible inter- and intratumoural heterogeneity between the primary tumour and the majority of metastatic sites.
* To map the natural history of the metastatic breast cancer process

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed active treatment (or trials) for metastatic breast cancer.
* Patients referred to either community or the hospital-based palliative care unit from Royal Marsden National Health Service Foundation Trust.

Exclusion Criteria:

* Lack of capacity / inability to give informed consent.
* Diagnosis of alternative cancer within the last 5 years other than resected basal cell skin cancer or cervical intraepithelial neoplasia.
* Patients known to be HIV, Hepatitis B virus or Hepatitis C virus positive on serology .
* Spongiform encephalopathy (known or suspected CJD) .
* Eligibility for or current participation in a clinical trial (excluding palliative care trials)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-09 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The acquisition of tumour tissue from multiple metastatic sites. | Within 6 hours from the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Barry, MB BS, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom